CLINICAL TRIAL: NCT06529510
Title: REThinkWELL- the Use of Therapeutic Game to Reduce Mental Health Symptoms in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REThinkWELL
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Emotional Problem; Mental Health Issue
Keywords: online therapeutic game; game-based CBT; emotional problems; mental health; children and adolescents
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REThink game (Experimental): Participants in this group will have access to the REThink therapeutic game for four weeks
  Interventions: Behavioral: REThink therpeutic game
- Care as usual (No Intervention): Participants in the control group do not receive an intervention but they have access to standard resources from the school

INTERVENTIONS:
Behavioral: REThink therpeutic game — REThink is an online therapeutic game aimed at enhancing the emotional health of young people, grounded in Rational Emotive Behavior Therapy (REBT). The game features a character named RETMAN, who guides players through seven levels, each focused on teaching a specific emotional regulation skill. Each level has three sub-levels that progressively increase in difficulty. REThink can be used as a standalone intervention, an adjunct to self-help psychotherapeutic approaches, or for targeted skills training.
  Arms: REThink game

SUMMARY:
To test the effect of a game-based intervention in reducing clinical and subclinical symptoms of children and adolescents.

DETAILED DESCRIPTION:
The general objective of the study is to test the REThink therapeutic game for improvements in clinical and subclinical mental health symptoms in children and adolescents aged 8-16 years old from multiple schools and counties. The game will be used by children and adolescents from the experimental group for a period of four weeks. Pre-test and post-test measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents aged 8 to 16 years
* subclinical level on the SDQ measure, total score, or emotional symptoms
* parental consent provided

Exclusion Criteria:

* intellectual disability or physical limitations precluding the use of the online game
* does not have parental informed consent

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 279 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Mental health | baseline assessment, one week prior to the intervention
  Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997). The scale has 25-items within its five subscales, namely emotional symptoms (ES), conduct problems (CP), hyperactivity/inattention (HY), peer relationship (PR) problems and prosocial behavior (PS) and total mental health difficulties score (MHD). The items are rated on a 3-point Likert scale, from 0 (not true) to 2 (certainly true). The minimum score is 0 and the maximum is 40. Higher scores represent higher level of mental health difficulties.
Changes in mental health | post-test assessment, one week after the intervention
  Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997). The scale has 25-items within its five subscales, namely emotional symptoms (ES), conduct problems (CP), hyperactivity/inattention (HY), peer relationship (PR) problems and prosocial behavior (PS) and total mental health difficulties score (MHD). The items are rated on a 3-point Likert scale, from 0 (not true) to 2 (certainly true). The minimum score is 0 and the maximum is 40. Higher scores represent higher level of mental health difficulties.
Irrationality | baseline assessment, one week prior to the intervention
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement"). The minimum score is 28 and the maximum score is 140. Higher scores represent higher levels of irrationality.
Changes in irrationality | post-test assessment, one week after the intervention
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement"). Higher scores represent higher levels of irrationality.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No